CLINICAL TRIAL: NCT03080129
Title: Microbiome and Sarcopenia in Patients With Liver Cirrhosis: A Prospective Controlled Cohort Study
Brief Title: Microbiome and Sarcopenia in Patients With Liver Cirrhosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SAR
Record Dates: First submitted 2017-03-01; First posted 2017-03-15 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Sarcopenia; Liver Cirrhosis
Keywords: Liver cirrhosis; Sarcopenia; Microbiome
MeSH Terms: conditions — Sarcopenia; Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cirrhosis + sarcopenia (Experimental): Patients with cirrhosis will receive 200ml of an oral nutritional supplement daily for 7 days.
  Interventions: Dietary Supplement: Fresubin energy
- Control (No Intervention): Patients with sarcopenia and no evidence of cirrhosis and healthy controls

INTERVENTIONS:
Dietary Supplement: Fresubin energy — dietary protein energy supplement
  Arms: Cirrhosis + sarcopenia

SUMMARY:
Protein-energy malnutrition (PEM) occurs in 65-90% of patients with liver cirrhosis. Severity of malnutrition correlates with progression of liver disease and leads to sarcopenia in 30-70% of cirrhotic patients. Malnutrition and sarcopenia are associated with an increased risk of complications and mortality.

In cirrhosis the gut microbiome is altered leading to increased gut permeability, bacterial translocation and inflammation. Since the microbiome is involved in nutrient uptake and metabolism, it is hypothesized that microbiome alterations contribute to sarcopenia. A prospective controlled cohort study to investigate the interrelation of microbiome changes and sarcopenia in cirrhosis will be conducted. Furthermore the effect of nutritional interventions on the microbiome in cirrhosis will be studied. From this study information on how the gut microbiome composition and sarcopenia are associated in cirrhosis and if modulation of the gut microbiome by nutritional interventions is feasible will be collected.

DETAILED DESCRIPTION:
Scientific background

Protein-energy malnutrition (PEM) occurs in 65-90% of patients with chronic liver disease. PEM is caused by various factors including poor dietary intake, loss of appetite, decreased hepatic protein synthesis, malabsorption and hypermetabolism. It is associated with an increased risk of complications including ascites, hepatic encephalopathy, variceal bleeding, hepatorenal syndrome and mortality. There is a direct relation between the progression of the liver disease and the severity of malnutrition.

Malnutrition and sarcopenia in liver cirrhosis patients

PEM leads to sarcopenia as a common, but frequently overlooked, complication. Sarcopenia is defined as a decrease in muscle mass two standard deviations below the healthy young adult mean. Sarcopenia is associated with aging, chronic diseases and malignancy. To determine the severity of muscle wasting, computed tomography scan (CT) or magnetic resonance imaging (MRI) are an objective and reproducible technique. Sarcopenia negatively impacts on survival, correlates with the risk of infections, increases surgical risk and leads to a poor quality of life. Besides PEM also inflammation is of importance in the development of sarcopenia.

Diversity in the microbiome in patients with liver cirrhosis and association with sarcopenia.

The gut microbiome of liver cirrhosis patients is altered compared to healthy individuals. Dysbiosis leads to an increased gut permeability, bacterial translocation and inflammation. This contributes to fibrogenesis and may also be related to hepatocarcinogenesis. Hence, new treatment approaches in cirrhosis focus on changing the microbial landscape.

Modulation the gut microbiome may also be a strategy to reverse sarcopenia by reducing systematic inflammation.

Hypothesis and aims

There is an association between gut microbiome composition, gut permeability and the existence of sarcopenia in cirrhotic patients.

Primary hypothesis: Diversity of the gut microbiome is reduced in liver cirrhosis patients with sarcopenia compared to those without sarcopenia or healthy controls.

Secondary hypotheses: There is an association between gut microbiome composition, biomarker of gut permeability and bacterial translocation with the presence of sarcopenia in cirrhosis. Oral nutrition supplements (ONS) can influence the composition of the gut microbiome, gut permeability, bacterial translocation and inflammation. Sarcopenia can be diagnosed from patients portraits.

Aims: to investigate:

* the composition of the gut microbiome
* biomarkers of gut permeability, bacterial translocation and inflammation
* the incidence and severity of sarcopenia
* the impact of oral nutrition supplements (ONS) on the gut microbiome
* whether artificial intelligence can be used to diagnose sarcopenia from face portraits.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients for any reason with clinical/radiological/histological diagnosis of cirrhosis
* Age >18y
* Informed consent
* CT/MRI scan within +/-14 days of the baseline study visit

Exclusion Criteria:

* Hepatic encephalopathy > grade 2 and or other cognitive disorder not allowing informed consent
* advanced hepatocellular carcinoma
* Any other condition or circumstance, which, in the opinion of the investigator, would affect the patient's ability to participate in the protocol

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Alpha diversity | day 1
  16s rDNA sequencing of the stool microbiome

SECONDARY OUTCOMES:
Zonulin | day 1
  ELISA
diamino-oxidase | day 1, day 7
  ELISA
Calprotectin | day 1
  ELISA
Gut permeability | change between day 1 and day 7
  marker panel
taxonomic composition of the microbiome | day 1
  16s rDNA sequencing of the stool microbiome
taxonomic composition of the microbiome | change between day 1 and day 7
  16s rDNA sequencing of the stool microbiome
lipopolysaccharide | day 1
  HEK blue cell assay
sCD14 | day 1
  ELISA
lipopolysaccharide binding protein | day 1
  ELISA
bacterial DNA | day 1
  HEK blue cell assay
bacterial translocation | change between day 1 and day 7
  marker panel
cytokine panel | day 1
  Bead array
carboxylated proteins | day 1
  ELISA
advanced oxidation end products | day 1
  ELISA
inflammation | change between day 1 and day 7
  marker panel
myostatin | day 1
  ELISA
fibroblast growth factor 21 | day 1
  ELISA
insulin like growth factor 1 | day 1
  ELISA
Irisin | day 1
  ELISA
nutritional status | day 1
  Questionnaire
Sarcopenia | day 1
  MR/CT scan
face portrait | day 1
  face portraits "selfies" will be obtained and AI algorithms will be used to diagnose sarcopenia from selfies

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Woltsche J, Pacher-Deutsch C, Furst S, Gulden L, Schwarzl J, Feldbacher N, Nepel M, Celcer L, Hasl N, Rieper V, Stadlbauer V, Horvath A. Microbial Dysbiosis in the Urinary Microbiome of Patients With Cirrhosis. Am J Gastroenterol. 2026 Jan 1;121(1):262-267. doi: 10.14309/ajg.0000000000003634. Epub 2025 Jul 7. PMID 40622440